CLINICAL TRIAL: NCT01805154
Title: Registry That Aims to Understand the Definition Used and Treatment Options Utilized by Clinicials for CRT Non-responders
Brief Title: Advance Cardiac Resynchronization Therapy (CRT) Registry
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 60046199
Record Dates: First submitted 2013-02-14; First posted 2013-03-06 (Estimated); Results first posted 2019-08-12 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CRT patients: Patients who have received any market approved St Jude Medical CRT-D or CRT-P device
  Interventions: Device: CRT Patients

INTERVENTIONS:
Device: CRT Patients — This is a group of patients who are receiving bi-ventricular pacing therapy from CRT device.
  Other Names: St Jude Medical, Any approved CRT device

SUMMARY:
The intent of this registry is to understand comprehensive clinical care strategies for Cardiac Resynchronization Therapy (CRT) patients especially non-responders in real-world clinical practice.

DETAILED DESCRIPTION:
Patients who are implanted CRT devices will be enrolled in the study. Once implanted, all patients will be followed at every 3 months for the first 12 months from the implant. The responder/non-responder evaluation will occur at 6 months from the implant date. The criteria used for determining the response to CRT will be captured.

During the office follow-up visits, arrhythmic episode diagnoses, device data and stored electrogram will be collected. All clinical events such as hospitalization for heart failure (HF), all-cause hospitalizations, and all-cause death will also be collected. For patients who are non-responders to CRT, any re-optimization of the device, i.e., atrioventricular and ventricle-to-ventricle interval optimization, left ventricular (LV) lead repositioning and pacing vector reconfiguration as well as modified/new clinical therapies administered in an attempt to improve HF condition will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Patient willing and able to sign informed consent
* Patients implanted with any market-approved St. Jude Medical CRT-D/P device with no prior LV lead placement

Exclusion Criteria:

* Are likely to undergo heart transplantation within the next 12 months
* Are less than 18 years of age
* Are pregnant or planning to become pregnant during the duration of the study
* Are currently participating in a clinical investigation that includes an active treatment arm
* Have a life expectancy of less than 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HF patients with St. Jude Medical CRT devices
Sampling Method: Probability Sample
Enrollment: 1529 (Actual)
Dates: Start 2013-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niraj Varma, MD, Study Chair — The Cleveland Clinic
Locations (69):
- United States (41):
  - Alabama Cardiovascular Group, P.C., Birmingham, Alabama
  - *Heart Center Research, LLC., Huntsville, Alabama
  - Cardiovascular Consultants Ltd, Glendale, Arizona
  - Cardiovascular Associates of Mesa, Mesa, Arizona
  - Phoenix Cardiovascular Research Group, Phoenix, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Comprehensive Cardiovascular, Bakersfield, California
  - Chula Vista Cardiac Center, Chula Vista, California
  - Cardiac Rhythm Specialist, Northridge, California
  - Claudio Bonometti MD, Inc, Santa Barbara, California
  - The Cardiac & Vascular Institute Research Foundation, LLC, Gainesville, Florida
  - Cardiology Consultants - Baptist Campus, Pensacola, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - VA Medical Center - Tampa, Tampa, Florida
  - Heartland Cardiovascular Center, Joliet, Illinois
  - Advocate Health and Hospitals Corporation, Oakbrook Terrace, Illinois
  - Unitypoint, Des Moines, Iowa
  - Heart Care Associates PSC, Madisonville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - St. Elizabeth's Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Cardiology Consultants of East Michigan, Flint, Michigan
  - *Thoracic Cardio Healthcare Found. (aka Sparrow Research), Lansing, Michigan
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Jackson Heart Clinic, Jackson, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - St. Louis University Hospital, St Louis, Missouri
  - Deborah Heart and Lung Center, Browns Mills, New Jersey
  - Lourdes Cardiology Services, Cherry Hill, New Jersey
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - Saint Vincent Consultants in Cardiovascular Diseases, Erie, Pennsylvania
  - Mountain States Medical Group Cardiology, Johnson City, Tennessee
  - Knoxville Cardiovascular Research Group, LLC, Knoxville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - North Texas Heart Center, Dallas, Texas
  - Martha Jefferson, Charlottesville, Virginia
  - University of Washington Medical Center, Seattle, Washington
  - Cardiac Rhythm Specialists, S.C., Milwaukee, Wisconsin
  - Cheyenne Cardiology Associates, Cheyenne, Wyoming
- Argentina (2):
  - Fundacion Favaloro para la Docencia e Inv. med., Buenos Aires, Riodepl
  - Instituto Cardiovascular Buenos Aires (ICBA), Buenos Aires, Riodepl
- Brazil (3):
  - Biocor Instituto, Nova Lima, Minas Gerais
  - Hospital Beneficiencia Portuguesa de Sao Paulo, São Paulo, Sao Pau
  - Instituto do Coracao (InCor) - HCFMUSP, São Paulo
- China (4):
  - Anhui Provincial Hospital, Hefei, Anhui
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - The First Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The 2nd Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang
- APEX Foundation, Medellín, Antioq, Colombia
- India (10):
  - Care Institute of Medical Sciences, Ahmedabad, Gujarat
  - Holy Family Hospital and Medical Research Center, Mumbai, Mhrshtr
  - Ruby Hall Clinic, Pune, Mhrshtr
  - Delhi Heart and Lung Institute, New Delhi, National Capital Territory of Delhi
  - Escorts Heart Institute and Research Centre, New Delhi, National Capital Territory of Delhi
  - Fortis Flt. Lt. Rajan Dhall Hospital, New Delhi, National Capital Territory of Delhi
  - Medanta - The Medicity Hospital, Gūrgaon, NCT DLH
  - Fortis Escorts Hospital, Amritsar, Punjab
  - Fortis Hospital, Mohali, Punjab
  - The Madras Medical Mission, Chennai, Tmlnadu
- Japan (4):
  - Fujita Health University School of medicine, Toyoake, Aichi-ken
  - Hirosaki University Hospital, Hirosaki-shi, Aomori
  - Kokura Memorial Hospital, Kitakyushu, Fukuoka
  - Chiba University, Chiba
- Heart Rhythm Management, San Juan, Puerto Rico
- South Korea (3):
  - Eulji university Hospital Daejeon, Daejeon, Hoseo
  - Samsung Medical Center, Seoul, Sudogwn
  - Yonsei University Health System, Seoul, Sudogwn

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Varma N, Wang JA, Jaswal A, Sethi KK, Kondo Y, Joung B, Yoo D, Auricchio A, Singh JP, Lee K, Gold MR. CRT Efficacy in "Mid-Range" QRS Duration Among Asians Contrasted to Non-Asians, and Influence of Height. JACC Clin Electrophysiol. 2022 Feb;8(2):211-221. doi: 10.1016/j.jacep.2021.09.012. Epub 2021 Nov 24. PMID 34838518
- [Derived] Varma N, Boehmer J, Bhargava K, Yoo D, Leonelli F, Costanzo M, Saxena A, Sun L, Gold MR, Singh J, Gill J, Auricchio A. Evaluation, Management, and Outcomes of Patients Poorly Responsive to Cardiac Resynchronization Device Therapy. J Am Coll Cardiol. 2019 Nov 26;74(21):2588-2603. doi: 10.1016/j.jacc.2019.09.043. PMID 31748196

RESULTS

PARTICIPANT FLOW:
Groups:
- Cardiac Resynchronization Therapy Patients: Patients who have received any market approved St Jude Medical cardiac resynchronization therapy defibrillator (CRT-D) or cardiac resynchronization therapy pacemaker (CRT-P) device.
  Cardiac resynchronization therapy patients: This is a group of patients who are receiving bi-ventricular pacing therapy from cardiac resynchronization therapy device.
Period: Overall Study
Arm/Group | Cardiac Resynchronization Therapy Patients
Started | 1529
Completed | 1175
Not Completed | 354

BASELINE CHARACTERISTICS:
Population: Of 1529 subjects enrolled, 5 were not included in baseline analyses (1 subject had incomplete informed consent and 4 did not have a device implant). Thus, only 1524 subjects were evaluable.
Groups:
- CRT Patients: Patients who have received any market approved St Jude Medical CRT-D or CRT-P device
  CRT Patients: This is a group of patients who are receiving bi-ventricular pacing therapy from a CRT device.
Arm/Group | CRT Patients
Number analyzed (Participants) | 1524
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 480
  Male | 1044
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Information was provided by 1428 subjects
  Participants
    Race/Ethnic category: number analyzed (Participants) | 1428
    Race/Ethnic category: American Indian or Alaska Native | 6
    Race/Ethnic category: Asian | 327
    Race/Ethnic category: Black or African American | 78
    Race/Ethnic category: Hispanic or Latino | 113
    Race/Ethnic category: White or Caucasian | 883
    Race/Ethnic category: Other | 21
Region of Enrollment [Number; unit: participants]
  Colombia | 27
  Argentina | 9
  United States | 1147
  India | 205
New York Heart Association (NYHA) Class [Count of Participants; unit: Participants] — NYHA Functional Classification has 4 categories:
  Class I (least severe) - no limitation of physical activity Class II - slight limitation of physical activity Class III - marked limitation of physical activity Class IV (most severe) - unable to carry on any physical activity without discomfort Population: information was available on 1522 subjects
  Participants
    number analyzed (Participants) | 1522
    NYHA Class I | 45
    NYHA Class II | 335
    NYHA Class III | 1033
    NYHA Class IV | 109
Type of Cardiomyopathy [Count of Participants; unit: Participants] — Population: Information was available on 1518 subjects
  Participants
    number analyzed (Participants) | 1518
    Ischemic | 597
    Non-Ischemic | 709
    None | 212
Left Ventricular Ejection Fraction % (EF) [Mean (Standard Deviation); unit: Percent blood ejected] — This is % of blood ejected from the left ventricle Population: Information was available on 1521 subjects
  Percent blood ejected
    number analyzed (Participants) | 1521
    (all) | 29.2 (11.2)
History of Atrial Fibrillation (AF) [Count of Participants; unit: Participants] — Population: Information was available on 1518 subjects
  Participants
    number analyzed (Participants) | 1518
    (all) | 583

OUTCOME MEASURES:

1. Primary Outcome: Number of CRT Non-responders Using 1) Clinical Composite Score (CCS) and 2) Site-specific Criteria for Determining CRT Response
Description: 1. The CCS has 4 components: New York Heart Association (NYHA) functional classification, Patient Global Assessment (PGA), heart failure (HF) events, cardiovascular death. NYHA Class ranges from Class I (least severe) to Class IV (most severe); possible PGA responses are "markedly worse", "moderately worse", "slightly worse", "no change", "slightly better", "moderately better, "markedly better". CCS components were used to classify or score subjects as "IMPROVED" (at least one-class improvement in NYHA Class or improvement by PGA "moderately" or "markedly" better AND no HF events AND no cardiovascular death), or "WORSENED" (worsening in NYHA Class OR worsening by PGA "moderately" or "markedly" worse OR presence of HF events OR Cardiovascular death, or "UNCHANGED" (neither "improved" or "worsened"). Note CCS is not a numeric score.
  2. Sites used their own clinical criteria (could include hospitalizations, functional assessments, etc.)
Time Frame: 6 months
Population: The analysis population included any subject who had a 6-month CRT evaluation or died due to a cardiovascular cause prior to 6 months. Subjects who withdrew prior to the 6-month visit, did not complete the 6-month visit or had relevant 6-month data missing were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Groups:
- CRT Patients: Patients who received any market approved St. Jude Medical CRT-D or CRT-P device.
Arm/Group | CRT Patients
Number analyzed (Participants) | 1327
Participants
  Site Determined CRT Response | 1061
  CCS Deteremined CRT Response | 900

2. Primary Outcome: Number of Subjects With Specfic Types of Symptom-based and Objective Definitions Used by Sites to Determine Patients' Response to CRT
Description: Number of subjects where sites used echocardiographic remodeling, clinical functional assessments, or clinical events to determine response status.
Time Frame: 6 months
Population: The analysis population included any subject with a completed 6-month CRT evaluation. Subjects who withdrew prior to the 6-month visit, did not complete the 6-month visit or had relevant 6-month data missing were excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | CRT Patients
Number analyzed (Participants) | 1299
Participants
  Echocardiographic Remodeling Used | 431
  Clinical Functional Assessment Used | 847
  Clinical Events Used | 858

3. Primary Outcome: Number of Subjects That Received Treatment Strategies for Heart Failure in the CRT Non-responder Population Between 6 and 12 Months
Time Frame: Between 6 and 12 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- CRT Patients: Patients who have received any market approved St. Jude Medical CRT-D or CRT-P device
Arm/Group | CRT Patients
Number analyzed (Participants) | 1299
Participants
  Device LV Pacing Change | 63
  Device AV/VV Intervals Optimized | 197
  Other Device Parameters Changed | 88
  Medication Changed | 319
  Arrythmia Treatments | 79
  Diet Compliance | 53
  Medication Compliance | 42
  HF Education Provided | 328
  Other Treatments | 71
  Treatment for Comorbidities | 100
  Bi-Ventricular Pacing Increase | 43

4. Primary Outcome: Number of Subjects Who Had an Improvement in NYHA Class Between Six Months and 12 Months
Description: Improvement in NYHA Class determined by improvement by at least 1 class.
Time Frame: Between 6 and 12 months
Population: Only subjects who had evaluable data at 6 and 12 months are included. Thus, fewer subjects than those who completed the 6-month and 12-month visits were analyzable.
Measure: Count of Participants; unit: Participants
Groups:
- Site CRT Responders: Patients who have received any market approved St Jude Medical CRT-D or CRT-P device
  CRT Patients: This is a group of patients who are receiving bi-ventricular pacing therapy from CRT device and were classified as CRT responders at 6 months.
- Site CRT Non-Responders: Patients who have received any market approved St Jude Medical CRT-D or CRT-P device
  CRT Patients: This is a group of patients who are receiving bi-ventricular pacing therapy from CRT device and were classified as CRT non-responders at 6 months.
Arm/Group | Site CRT Responders | Site CRT Non-Responders
Number analyzed (Participants) | 559 | 90
Participants | 93 | 34

ADVERSE EVENTS:
Time Frame: Data were collected and reported over the 12-month study period.
Groups:
- CRT Patients: Patients who have received any market approved St Jude Medical CRT-D or CRT-P device CRT Patients: This is a group of patients who are receiving bi-ventricular pacing therapy from CRT device.
  Of 1529 subjects enrolled, 5 were not included in analysis (1 had incomplete informed consent and 4 did not receive a device implant).
Arm/Group | CRT Patients
All-Cause Mortality (participants affected / at risk) | 132/1524
Serious Adverse Events (participants affected / at risk) | 226/1524
Other Adverse Events (participants affected / at risk) | 403/1524
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT Patients (N=1524)
Acute CHF (Cardiac disorders) | 70 (102)
Atrial Arrythmia (Cardiac disorders) | 12 (14)
Atrial Fib Ablation (Cardiac disorders) | 3 (3)
Air Embolism (Injury, poisoning and procedural complications) | 1 (1)
Arrest Cardiopulmonary (Injury, poisoning and procedural complications) | 4 (4)
BLEEDING(NON-HEMATOMA) (Injury, poisoning and procedural complications) | 7 (7)
CARDIAC TAMPONADE (Injury, poisoning and procedural complications) | 2 (2)
CARDIAC/CORONARY SINUS DISSECTION (Injury, poisoning and procedural complications) | 1 (1)
CHEST PAIN (Cardiac disorders) | 1 (1)
ER VISIT AND OBSERVATION ADMISSION (Injury, poisoning and procedural complications) | 1 (1)
EROSION/EXTRUSION (Infections and infestations) | 3 (3)
HEMATOMA (Injury, poisoning and procedural complications) | 6 (7)
HOSPITALIZATION FOR DECREASED MENTAL STATUS AND FEVER (General disorders) | 1 (1)
INFECTION (Infections and infestations) | 7 (7)
LEAD DISLODGEMENT OR MIGRATION (Injury, poisoning and procedural complications) | 41 (51)
RA LEAD FRACTURE (Product Issues) | 1 (1)
RV LEAD MALFUNCTION (Product Issues) | 1 (1)
LV LOSS OF CAPTURE (Product Issues) | 2 (3)
MYOCARDIAL INFARCTION (Cardiac disorders) | 19 (20)
NEW OR WORSENED ANGINA (Cardiac disorders) | 4 (4)
OTHER Cardiac (Cardiac disorders) | 8 (10)
OTHER Death (Cardiac disorders) | 5 (5)
OTHER Gastro (Gastrointestinal disorders) | 6 (6)
OTHER General (General disorders) | 37 (43)
OTHER Infections (Infections and infestations) | 14 (17)
Other Respiratory (Respiratory, thoracic and mediastinal disorders) | 7 (11)
PERICARDIAL EFFUSION (Injury, poisoning and procedural complications) | 2 (2)
PHRENIC NERVE/DIAPHRAGMATIC STIMULATION (Injury, poisoning and procedural complications) | 2 (2)
PNEUMOTHORAX (Injury, poisoning and procedural complications) | 3 (3)
SOB; EDEMA; DIURESIS; MONITORING (General disorders) | 1 (1)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULSE GENERATOR MALFUNCTION (Product Issues) | 1 (1)
SHOCK/HYPOTENSION (Injury, poisoning and procedural complications) | 5 (6)
SYNCOPE UNKNOWN ETIOLOGY (General disorders) | 2 (2)
THROMBO-EMBOLIC EVENT (General disorders) | 2 (2)
TRIMALLEOLAR FRACTURE RIGHT ANKLE (Musculoskeletal and connective tissue disorders) | 1 (1)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 11 (11)
WORSENING CAD (Cardiac disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CRT Patients (N=1524)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1)
ARREST - CARDIOPULMONARY (Cardiac disorders) | 2 (2)
ASYSTOLE (Cardiac disorders) | 1 (1)
ATRIAL ARRHYTHMIA (Cardiac disorders) | 37 (39)
BLEEDING(NON-HEMATOMA) (Injury, poisoning and procedural complications) | 7 (7)
CHEST PAIN (General disorders) | 1 (1)
CLOSTRIDIUM DIAARHEA (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1)
DECOMPENSATED HF (Cardiac disorders) | 98 (133)
DIZZINESS, NAUSEA, IRREGULAR HEART BEAT (General disorders) | 1 (1)
ELEVATED PACING THRESHOLDS (Product Issues) | 14 (14)
FATIGUE (General disorders) | 1 (1)
HEART FAILURE (Cardiac disorders) | 1 (1)
HEMATOMA (Injury, poisoning and procedural complications) | 17 (18)
HEMOTHORAX (Injury, poisoning and procedural complications) | 1 (1)
HIGH DFT'S (Product Issues) | 1 (1)
INFECTION (Infections and infestations) | 25 (26)
LEAD DISLODGEMENT OR MIGRATION (Injury, poisoning and procedural complications) | 5 (5)
Lead Noise (Product Issues) | 3 (3)
LOSS OF CAPTURE (Product Issues) | 6 (7)
LOSS OF SENSING (Product Issues) | 2 (2)
LOW CARDIAC OUTPUT SYNDROME AND PULMONARY OEDEMA (Cardiac disorders) | 1 (1)
LOWER EXTREMITY EDEMA (Vascular disorders) | 1 (1)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
NEW OR WORSENED ANGINA (Cardiac disorders) | 7 (7)
OTHER Cardiac (Cardiac disorders) | 18 (20)
OTHER Gastro (Gastrointestinal disorders) | 26 (26)
OTHER General (General disorders) | 174 (284)
OTHER Implant (Injury, poisoning and procedural complications) | 12 (12)
OTHER Infections (Infections and infestations) | 37 (53)
Other Respiratory (Respiratory, thoracic and mediastinal disorders) | 18 (23)
OVERSENSING (Product Issues) | 9 (10)
OVERSENSING RESULTING IN THERAPY (Product Issues) | 1 (1)
PACEMAKER MEDIATED TACHYCARDIA (PMT) (Product Issues) | 5 (5)
PERICARDIAL EFFUSION (Injury, poisoning and procedural complications) | 2 (2)
PHRENIC NERVE/DIAPHRAGMATIC STIMULATION (Product Issues) | 33 (38)
PNEUMOTHORAX (Injury, poisoning and procedural complications) | 1 (1)
SHOCK/HYPOTENSION (Infections and infestations) | 5 (5)
SYNCOPE UNKNOWN ETIOLOGY (General disorders) | 7 (7)
THERAPY FOR NON-VENTRICULAR RHYTHM (Cardiac disorders) | 9 (13)
THROMBO-EMBOLIC EVENT (General disorders) | 6 (6)
UNDERSENSING (Product Issues) | 2 (2)
UPPER RESIRATORY TRACT INFECTION (Infections and infestations) | 1 (1)
VENTRICULAR ARRHYTHMIA (Cardiac disorders) | 7 (51)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2015-12-17): https://cdn.clinicaltrials.gov/large-docs/54/NCT01805154/Prot_ICF_000.pdf